CLINICAL TRIAL: NCT03897569
Title: Association Between Ankle Dorsiflexion and Frontal Projection Angle During a Functional Task in the Patellofemoral Pain Syndrome
Brief Title: Association Between Ankle Dorsiflexion and Frontal Projection Angle in PFPS
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Karima Abdelaty Hassan, principal investigator, Cairo University
Other Study IDs: PFPS kinematics
Record Dates: First submitted 2019-03-27; First posted 2019-04-01 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: Patellofemoral Pain Syndrome; knee kinematics; frontal projection angle; ankle motion
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- patellofemoral pain syndrome: twenty subjects with anterior or retropatellar knee pain from at least 2 of the following Activities : (1) prolonged sitting; (2) stair climbing; (3) squatting; (4) running; (5) kneeling; and (6) hopping/jumping.
  Interventions: Other: frontal projection angle, ankle dorsiflexion
- control: twenty-six asymptomatic subject will be recruited for this study and should have no pain or other relevant clinical symptoms in the lower quadrant
  Interventions: Other: frontal projection angle, ankle dorsiflexion

INTERVENTIONS:
Other: frontal projection angle, ankle dorsiflexion — Dorsiflexion measurements will be taken in 4 different positions and repeated and recorded 3 times in each position, Prone bent, straight knee and Standing bent, straight knee. Prior to the measurement, the participants completed two 30-second calf stretches The FPPA was determined as the angle at the knee formed by lines connecting the anterior superior iliac spine, the midpoint of the femoral condyles and the midpoint of the malleoli at the deepest part of the squat

SUMMARY:
The study will investigate an association between ankle dorsiflexion and altered frontal knee kinematics during step down test in patients with PFPS.

DETAILED DESCRIPTION:
Altered frontal and transverse plane hip kinematics during single leg weight-bearing tasks are thought to be important contributors to patellofemoral pain (PFP). The closed chain nature of single leg tasks means that hip kinematics can be influenced by more distal mechanics, such as foot pronation.

One of the often-studied distal movements theorized to cause PFPS is pronation of the subtalar joint. Pronation is a tri-planar movement that includes dorsiflexion, eversion, and abduction of the foot. Many studies have examined eversion characteristics of PFPS patients, but the dorsiflexion aspect of the movement has been shown to be a possible risk factor, restricting dorsiflexion was shown to increase medial knee displacement in young healthy adults. Conversely, when available dorsiflexion ROM is increased, medial knee displacement is thought to decrease.

Patients with PFPS were observed to have a decreased DFROM (dorsiflexion range of motion) as compared to normal individuals, though this topic has not thoroughly been investigated.

ELIGIBILITY:
Inclusion Criteria:

1. Anterior or retropatellar knee pain from at least 2 of the following Activities : (1) prolonged sitting; (2) stair climbing; (3) squatting; (4) running; (5) kneeling; and (6) hopping/jumping.
2. Insidious onset of symptoms unrelated to a traumatic incident and persistent for at least 6weeks.
3. VAS equal to or greater than 3.
4. Age of the subject 18-35 years to limit the possibility that PFPS over age 35 may have been complicated by arthritic changes, and also the subjects should have closed epiphyseal growth plates.
5. BMI under 30 kg/m2, both gender

For the control group, subjects were recruited to this study if they had:

1. No previous history or diagnosis of knee pathology.
2. No pain with any of the above-mentioned provocative activities.
3. No history of lower limb or spinal pathology.

Exclusion Criteria:

1. A history of any of the following condition: meniscal or other intraarticular pathologic conditions; cruciate or collateral ligament involvement.
2. A history of traumatic patellar subluxation or dislocation.
3. Previous surgery in the lower extremities within the 12 months prior to participation in the study.
4. Any balance impairments are secondary to a vestibular or neurological disorder or secondary to the use of medication.
5. Any lower limb bony/congenital deformity

Ages: 18 Years to 35 Years | Sex: All
Age Groups: Adult
Study Population: Subjects between 18 to 35 years old with symptomatic patellofemoral pain syndrome and healthy control.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2019-03-30 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Frontal knee kinematic | 20 minutes
  The knee kinematic will be measured by using digital video camera using single leg squat during functional step down test

SECONDARY OUTCOMES:
Ankle mobility | 20 minutes
  Ankle dorsiflexion ROM will be assessed by bubble inclinometer during weight-bearing and non-weight-bearing positions.

CONTACTS AND LOCATIONS:
Overall Officials: karima A Hassan, PhD, Principal Investigator — Cairo University
Locations (1):
- Faculty of Physical therapy, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No